CLINICAL TRIAL: NCT00878657
Title: Phase I/II Radiotherapy Dose Escalation Study in Locally Advanced Pancreatic Cancer, Using a Simultaneous Intensity Modulated Boost With Concurrent Gemcitabine
Brief Title: Intensity-Modulated Radiation Therapy and Gemcitabine in Treating Patients With Locally Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000639635; P30CA072720 (NIH); CINJ-070805 (Other: Rutgers Cancer Institute of New Jersey); 0220090024 (Other: The Rutgers RBHS Institutional Review Board)
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy plus gemcitabine (Experimental): Drug: gemcitabine hydrochloride
  Radiation: intensity-modulated radiation therapy
  Interventions: Drug: gemcitabine hydrochloride; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Pre-Chemoradiation (Induction) Chemotherapy Gemcitabine will be given weekly for seven doses at a dose of 1000 mg/m2/wk (Days 1, 8, 15, 22, 29, 36, 43) unless toxicity develops. Chemoradiation gemcitabine will be given 400 mg/m2, infused over 30 minutes, within 120 minutes before radiotherapy. Post-chemoradiation chemotherapy, patients will receive two cycles of gemcitabine. A cycle will be defined as three weeks of gemcitabine at 1000 mg/m2/d, once weekly, followed by a one-week rest.
Radiation: intensity-modulated radiation therapy — Dose escalation levels (cohorts) for this study:
  Dose Level 1: GTV plus drainage areas 45 Gy, Boost GTV 50.4 Gy Dose Level 2: GTV plus drainage areas 45 Gy, Boost GTV 54.0 Gy Dose Level 3: GTV plus drainage areas 45 Gy, Boost GTV 59.4 Gy Dose Level 4: GTV plus drainage areas 45 Gy, Boost GTV 64.8 Gy Dose Level 5: GTV plus drainage areas 45 Gy, Boost GTV 70.2 Gy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving intensity-modulated radiation therapy together with gemcitabine may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of intensity-modulated radiation therapy and to see how well it works when given together with gemcitabine in treating patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
The study was terminated early due to slow accrual and only the phase I portion of hte study was opened. The phase of the study has been revised to only a phase I study.

OBJECTIVES:

* To determine the maximum tolerated dose (MTD) of intensity-modulated radiotherapy delivered to the gross tumor volume when administered with gemcitabine hydrochloride in patients with locally advanced pancreatic carcinoma. (Phase I)
* To define the dose-limiting toxicities of this regimen in these patients. (Phase I)
* To determine the local control in patients treated at the MTD (determined in phase I). (Phase II)
* To compare the disease-free survival and time to progression in these patients with that of historical controls. (Phase II)

OUTLINE: This is a multicenter phase I, dose-escalation study of intensity-modulated radiotherapy, followed by a phase II study.

* Induction chemotherapy: Patients receive gemcitabine hydrochloride IV on days 1, 8, and 15. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo CT scan. Patients with no evidence of metastatic disease proceed to chemoradiotherapy.
* Chemoradiotherapy: Beginning 1-2 weeks after completion of induction chemotherapy, patients undergo intensity-modulated radiotherapy once daily 5 days a week and gemcitabine hydrochloride IV over 30 minutes once weekly for 5 weeks in the absence of disease progression or unacceptable toxicity. Patients whose disease remains unresectable proceed to adjuvant chemotherapy.
* Adjuvant chemotherapy: Beginning 4-6 weeks after completion of chemoradiotherapy, patients receive gemcitabine hydrochloride as in induction chemotherapy.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed adenocarcinoma or poorly differentiated carcinoma of the pancreas, ampulla of Vater, or distal bile duct

  * Locally advanced disease
  * Medically inoperable, unresectable, or borderline resectable disease

    * No previously resected disease (i.e., status post-pancreaticoduodenotomy)
* No non-adenocarcinoma, adenosquamous carcinoma, islet cell carcinoma, cyst adenoma, cystadenocarcinoma, carcinoid tumor, or duodenal carcinoma
* No lesions in the tail of the pancreas and/or splenic artery/vein involvement/encasement
* No recurrent or metastatic (M1) disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* WBC > 3,000/μL
* Platelet count > 100,000/μL
* Bilirubin ≤ 2 mg/dL
* SGOT < 5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate oral nutrition (e.g., ≥ 1,500 calories/day, stable weight for ≥ 2 weeks, and ≤ 5% weight loss)
* No active malignancy within the past 3 years, except cervical carcinoma in situ or nonmelanoma skin cancer that has been removed
* No severe, active comorbidity, including any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring IV antibiotics at the time of study registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization within the past month or precluding study therapy at the time of study registration
  * Active hepatitis, decompensated cirrhosis, or clinically significant liver failure
  * Other severe comorbid condition, as determined by the principal investigator

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy
* No prior radiotherapy to any upper abdominal site
* No concurrent prophylactic colony-stimulating factors during radiotherapy
* No concurrent warfarin
* No other concurrent chemotherapy, immunotherapy, hormonal cancer therapy, radiotherapy, surgery for cancer, or experimental therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-04; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of intensity-modulated radiotherapy (Phase I) | 4 years
Overall survival (Phase II) | 4 years
Disease-free survival (Phase II) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Salma Jabbour, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States